CLINICAL TRIAL: NCT00433550
Title: A Phase II Trial of Pharmacogenetic-Based Dosing of Irinotecan, Oxaliplatin, and Capecitabine as First-Line Therapy for Advanced Small Bowel Adenocarcinoma
Brief Title: Irinotecan, Oxaliplatin, and Capecitabine as First-Line Therapy in Treating Patients With Metastatic or Unresectable Locally Advanced Small Bowel Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0543; NCI-2009-00650 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000528263 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Small Intestine Adenocarcinoma; Recurrent Small Intestine Cancer
MeSH Terms: interventions — Capecitabine; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (6/6 UGT1A1 genotype) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes and oxaliplatin IV over 2 hours on day 1 and capecitabine PO BID on days 2-15
  Interventions: Drug: capecitabine; Drug: irinotecan hydrochloride; Drug: oxaliplatin
- Group 2 (6/7 UGT1A1 genotype) (Experimental): Patients receive irinotecan hydrochloride as in group 1. They also receive oxaliplatin and capecitabine as in group 1 but at lower doses.
  Interventions: Drug: capecitabine; Drug: irinotecan hydrochloride; Drug: oxaliplatin
- Group 3 (7/7 UGT1A1 genotype) (Experimental): Patients receive irinotecan hydrochloride, oxaliplatin, and capecitabine as in group 1 but at lower doses.
  Interventions: Drug: capecitabine; Drug: irinotecan hydrochloride; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine — given orally
Drug: irinotecan hydrochloride — given IV
Drug: oxaliplatin — given IV

SUMMARY:
This phase II trial studies how well giving irinotecan hydrochloride together with oxaliplatin and capecitabine works as first-line therapy in treating patients with metastatic or unresectable locally advanced small bowel cancer. Drugs used in chemotherapy, such as irinotecan hydrochloride, oxaliplatin, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To assess the confirmed tumor response of the combination of oxaliplatin, irinotecan (irinotecan hydrochloride), and capecitabine in patients with advanced adenocarcinoma of the small bowel when dosed according to UGT1A1 genotype.

SECONDARY OBJECTIVES:

1. To assess the toxicity of this regimen in these groups of patients.
2. To gain preliminary data on whether microsatellite instability influences outcome within this arm.
3. To gain preliminary data on whether evidence of celiac disease may affect toxicity and outcome.
4. To gain preliminary data on whether site of tumor origin (duodenal, jejunal, or ileal) affects response or survival.

OUTLINE: Patients are assigned to 1 of 3 treatment groups based on UGT1A1 genotype.

GROUP 1 (6/6 UGT1A1 genotype): Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes and oxaliplatin IV over 2 hours on day 1 and capecitabine orally (PO) twice daily (BID) on days 2-15.

GROUP 2 (6/7 UGT1A1 genotype): Patients receive irinotecan hydrochloride as in group 1. They also receive oxaliplatin and capecitabine as in group 1 but at lower doses.

GROUP 3 (7/7 UGT1A1 genotype): Patients receive irinotecan hydrochloride, oxaliplatin, and capecitabine as in group 1 but at lower doses.

In all groups, treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After the completion of study treatment, patients are followed every 6 weeks for 2 years and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria

* Confirmation UDP glucuronosyltransferase 1 family, polypeptide A complex locus (UGT1A1) TA indel genotype of 6/6, 6/7, or 7/7 after pre-registration but prior to registration
* Patient willingness to provide a serum sample for analysis for celiac disease (tissue transglutaminase antibodies)
* Small bowel adenocarcinoma, either metastatic or locally advanced and not surgically resectable; NOTE: periampullary carcinoma and appendiceal cancer are not eligible
* Histologic or cytologic confirmation of adenocarcinoma consistent with small bowel origin; biopsy can be of primary tumor or can be from a metastatic site if there is a primary small bowel tumor currently or previously present
* Measurable disease; for patients with lesions >= 1 cm but < 2 cm, spiral computed tomography (CT) scan imaging must be used for tumor assessments
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* >= 4 weeks since prior major surgery to time of registration
* >= 2 weeks from completion of any radiation treatment
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Serum glutamic oxaloacetic transaminase (SGOT) =< 5 x upper normal limit (UNL); =< 2.5 x UNL if no liver metastases
* Total bilirubin:

  * For 6/6 patients: =< upper limit of normal (ULN)
  * For 6/7 or 7/7 patients: =< 2.0 x ULN
* Hemoglobin >= 9.0 g/dL
* Creatinine =< 1.5 x UNL (if > 1.5 x UNL, calculated creatinine clearance should be checked.; if it is > 60 mL/min, then the patient is eligible for the study)
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

Exclusion Criteria

* Prior chemotherapy regimen for advanced small bowel cancer (prior adjuvant chemotherapy with fluorouracil (5FU)/leucovorin is permitted if last dose was administered >= 3 months prior to registration); prior oxaliplatin or irinotecan use as adjuvant therapy is not permitted
* Prior radiotherapy to > 25% of bone marrow
* Active or uncontrolled infection
* Evidence of serious intercurrent illness (e.g., unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia)
* Pregnant women; women of child-bearing potential and men must agree to use adequate contraception (diaphragm, birth control pills, injections, foams, intrauterine device [IUD], or abstinence, etc.) for the duration of study participation; if a woman becomes pregnant or suspects that she is pregnant while participating in this study, she should inform her treating physician immediately and all study treatment discontinued
* Nursing women; breast-feeding should be discontinued when the mother is treated with these agents
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Current evidence of other malignancy besides small bowel adenocarcinoma, with exception of non-melanoma skin cancer
* Known central nervous system metastases or carcinomatous meningitis
* Preexisting sensory neuropathy >= grade 2 from any cause interfering with function
* Concurrent therapy with sorivudine, brivudine, lamivudine, or stavudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-05; Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McWilliams, MD, Study Chair — Mayo Clinic
Locations (115):
- United States (115):
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Derived] Goetz MP, McKean HA, Reid JM, Mandrekar SJ, Tan AD, Kuffel MA, Safgren SL, McGovern RM, Goldberg RM, Grothey AA, McWilliams R, Erlichman C, Ames MM. UGT1A1 genotype-guided phase I study of irinotecan, oxaliplatin, and capecitabine. Invest New Drugs. 2013 Dec;31(6):1559-67. doi: 10.1007/s10637-013-0034-9. Epub 2013 Oct 10. PMID 24114122

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to registration, patients were tested for UGT1A1 TA indel genotype of 6/6, 6/7, or 7/7. Patients were grouped into one of three treatment groups depending on UGT1A1 genotype. All other genotypes were ineligible. The endpoints of this study are not to compare results between the UGT1A1 types, but to analyze as one combined cohort.
Groups:
- Group 1 (6/6 UGT1A1 Genotype): Patients receive 150 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 100 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 1600 mg/m^2/day capecitabine PO BID on days 2-15
- Group 2 (6/7 UGT1A1 Genotype): Patients receive 150 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 400 mg/m^2/day capecitabine PO BID on days 2-15
- Group 3 (7/7 UGT1A1 Genotype): Patients receive 75 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 400 mg/m^2/day capecitabine PO BID on days 2-15
Period: Overall Study
Arm/Group | Group 1 (6/6 UGT1A1 Genotype) | Group 2 (6/7 UGT1A1 Genotype) | Group 3 (7/7 UGT1A1 Genotype)
Started | 17 | 10 | 6
Completed | 17 | 10 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients registered were analyzed for baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (6/6 UGT1A1 Genotype) | Group 2 (6/7 UGT1A1 Genotype) | Group 3 (7/7 UGT1A1 Genotype) | Total
Number analyzed (Participants) | 17 | 10 | 6 | 33
Age, Continuous [Median (Full Range); unit: years] | 64 [41 to 75] | 66.5 [42 to 77] | 62.5 [43 to 74] | 64 [41 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 9
  Male | 12 | 9 | 3 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 10 | 6 | 33

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Tumor Response Rate (Proportion of Participants With Complete Response)
Description: Evaluated using RECIST version 1.0. Confirmed tumor response rate was defined as achieving partial response (PR) or complete response (CR) in two consecutive assessments at least 6 weeks apart. CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. The confirmed response rate is reported as the number of participants with confirmed responses divided by the number of evaluated participants.
Time Frame: 36 weeks
Population: One patient was later found to be a major treatment violation during cycle 1 and was not included in this analysis. All the other 32 patients were analyzed together for this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Groups:
- All Patients (6/6, 6/7, 7/7 UGT1A1 Genotype): Group 1 (6/6 UGT1A1 genotype):
  Patients receive 150 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 100 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 1600 mg/m^2/day capecitabine PO BID on days 2-15
  Group 2 (6/7 UGT1A1 genotype):
  Patients receive 150 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 400 mg/m^2/day capecitabine PO BID on days 2-15.
  Group 3 (7/7 UGT1A1 genotype):
  Patients receive 75 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 400 mg/m^2/day capecitabine PO BID on days 2-15
Arm/Group | All Patients (6/6, 6/7, 7/7 UGT1A1 Genotype)
Number analyzed (Participants) | 32
proportion of patients | .38 [.21 to .56]

2. Secondary Outcome: Overall Survival
Description: Overall survival will be defined as the time from registration to death. Patients lost to follow-up for this endpoint will be censored at the date of last contact (i.e., last known alive). The distribution of overall survival will be estimated using Kaplan-Meier methodology.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Patients (6/6, 6/7, 7/7 UGT1A1 Genotype): Group 1 (6/6 UGT1A1 genotype):> Patients receive 150 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 100 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 1600 mg/m^2/day capecitabine PO BID on days 2-15> > Group 2 (6/7 UGT1A1 genotype):> Patients receive 150 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 400 mg/m^2/day capecitabine PO BID on days 2-15.>
  > Group 3 (7/7 UGT1A1 genotype):> Patients receive 75 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 400 mg/m^2/day capecitabine PO BID on days 2-15
Arm/Group | All Patients (6/6, 6/7, 7/7 UGT1A1 Genotype)
Number analyzed (Participants) | 32
months | 13.4 [10.5 to 18.1]

3. Secondary Outcome: Progression Free Survival
Description: Time to disease progression is defined as the time from registration to the earlier of documentation of disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The distribution of time to progression will be estimated using Kaplan-Meier methodology.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Patients (6/6, 6/7, 7/7 UGT1A1 Genotype): Group 1 (6/6 UGT1A1 genotype):
  > Patients receive 150 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 100 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 1600 mg/m^2/day capecitabine PO BID on days 2-15
  >
  >
  Group 2 (6/7 UGT1A1 genotype):
  > Patients receive 150 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 400 mg/m^2/day capecitabine PO BID on days 2-15.
  >
  >
  Group 3 (7/7 UGT1A1 genotype):
  > Patients receive 75 mg/m^2 irinotecan hydrochloride IV over 90 minutes and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 400 mg/m^2/day capecitabine PO BID on days 2-15
Arm/Group | All Patients (6/6, 6/7, 7/7 UGT1A1 Genotype)
Number analyzed (Participants) | 32
months | 8.9 [4.7 to 10.8]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented. Duration of response will be analyzed using Kaplan-Meier methods.
Time Frame: Up to 2 years
Population: All patients who achieved a CR or PR are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients (6/6, 6/7, 7/7 UGT1A1 Genotype)
Number analyzed (Participants) | 12
months | 9.0 [7.8 to NA] — Too few events have occurred to estimate the upper 95% Confidence Interval.

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from the date of registration to the date at which the patient is removed from treatment due to progression, toxicity, or refusal. If the patient is considered to have had a major treatment violation or is taken off study as a non-protocol failure, the patient will be censored on the date they are removed from treatment. Time to treatment failure will be analyzed using Kaplan-Meier methods.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients (6/6, 6/7, 7/7 UGT1A1 Genotype)
Number analyzed (Participants) | 32
months | 6.7 [4.3 to 10.6]

ADVERSE EVENTS:
Arm/Group | Group 1 (6/6 UGT1A1 Genotype) | Group 2 (6/7 UGT1A1 Genotype) | Group 3 (7/7 UGT1A1 Genotype)
Serious Adverse Events (participants affected / at risk) | 7/17 | 6/10 | 1/6
Other Adverse Events (participants affected / at risk) | 16/17 | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (6/6 UGT1A1 Genotype) (N=17) | Group 2 (6/7 UGT1A1 Genotype) (N=10) | Group 3 (7/7 UGT1A1 Genotype) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (6) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 3 (5) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (6) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (6/6 UGT1A1 Genotype) (N=17) | Group 2 (6/7 UGT1A1 Genotype) (N=10) | Group 3 (7/7 UGT1A1 Genotype) (N=6)
Hemoglobin decreased (Blood and lymphatic system disorders) | 13 (120) | 10 (58) | 6 (57)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Eye disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 16 (66) | 7 (25) | 4 (19)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Esophageal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (4) | 4 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (71) | 7 (31) | 6 (20)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (39) | 4 (13) | 6 (16)
Fatigue (General disorders) | 5 (10) | 6 (16) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (2) | 0 (0)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 11 (45) | 7 (26) | 3 (16)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 10 (39) | 7 (26) | 3 (13)
Platelet count decreased (Investigations) | 11 (48) | 5 (9) | 1 (17)
Weight loss (Investigations) | 2 (2) | 1 (3) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal (Nervous system disorders) | 3 (9) | 2 (9) | 1 (5)
Memory impairment (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (98) | 7 (41) | 5 (33)
Taste alteration (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (13) | 5 (13) | 1 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 2 (6) | 1 (9)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (81) | 9 (53) | 5 (51)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 7 (11) | 2 (4) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less